CLINICAL TRIAL: NCT07224035
Title: Helicobacter Pylori Screening and Treatment in the At-risk South Florida Community- AIM 1
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Phathom Pharmaceuticals (Unknown); NRG Oncology (Other)
Responsible Party: Principal Investigator, Shria Kumar, Assistant Professor of Clinical Medicine, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20211207-AIM 1
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: H Pylori Infection; H Pylori Gastritis; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Helicobacter Pylori Screening and Treatment (Experimental): Participants in this single-arm study will undergo screening for Helicobacter pylori (H. pylori) using the PYtest® 14C-Urea Capsule Breath Test. This FDA-approved, non-invasive diagnostic method involves swallowing a radiolabeled urea capsule. If gastric urease from H. pylori is present, the urea is hydrolyzed to produce carbon dioxide and ammonia. Ten minutes after ingestion, a breath sample is collected in a balloon and transferred into a collection fluid to trap the labeled carbon dioxide. The sample is analyzed using a liquid scintillation counter to determine infection status.
  Participants who test positive will receive VOQUEZNA® Triple Pak® therapy, dispensed by the study team at the time of diagnosis. Phathom Pharmaceuticals will supply the medications (which include complete medication package insert), but the study team hold and dispenses medications.
  Interventions: Drug: PYTEST® 14C-Urea Breath Test; Drug: VOQUEZNA® Triple Pak®

INTERVENTIONS:
Drug: PYTEST® 14C-Urea Breath Test — FDA-approved radiolabeled urea capsule used in the PYtest® 14C-Urea Breath Test for non-invasive detection of H. pylori. Participants ingest the capsule, and breath samples are collected and analyzed to determine infection status.
Drug: VOQUEZNA® Triple Pak® — FDA-approved combination therapy for H. pylori infection, consisting of:
  Vonoprazan tablets 20 mg (1 tablet twice daily for 14 days) Amoxicillin 500 mg (2 tablets twice daily for 14 days) Clarithromycin 500 mg (1 tablet twice daily for 14 days) Medications are dispensed by the study team at the time of diagnosis.

SUMMARY:
H. pylori is an infection of the stomach that can cause chronic gastritis, gastric cancer and peptic ulcer disease. The goal of this study is to screen people for this infection and offer treatment for those who test positive for the infection. By treating those who are positive for H. pylori, there is an opportunity to prevent gastritis, peptic ulcer disease, and even gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age

Exclusion Criteria:

* Adults with a personal history of gastric cancer
* Adults with prior history of H. Pylori (HP) treatment and confirmed eradication
* Adults unable to consent
* Adults unable to consent in their preferred language
* Pregnant women, those who are breastfeeding, or those who are planning to become pregnant/breastfeed
* Prisoners
* Persons who are allergic, hypersensitive, or unable to take any of the components of the medication regimen VOQUEZNA® Triple Pak®:
* vonoprazan
* amoxicillin or any other beta-lactams (e.g. penicillins and cephalosporins)
* clarithromycin or any other macrolide antimicrobial (e.g. erythromycin)
* Persons presently taking any of the following:
* Rilpivirine-containing products
* Pimozide
* Lomitapide, lovastatin, simvastatin, atorvastatin, and pravastatin
* Ergot alkaloids
* Colchicine (if with kidney or liver impairment)
* Lurasidone
* Drugs known to prolong the QT interval (e.g., pimozide).
* Class IA (e.g., quinidine, procainamide, disopyramide) or Class III (e.g., dofetilide, amiodarone, sotalol) antiarrhythmic agents
* Verapamil, amlodipine, diltiazem, nifedipine
* Nateglinide, pioglitazone, repaglinide, rosiglitazone, and insulin
* Quetiapine
* Warfarin
* Benzodiazepines (e.g. triazolam, midazolam)
* Persons who have any of the following, as they may be prone to adverse effects from the medication regimen:
* History of cholestatic jaundice
* Severe kidney impairment
* Severe hepatic impairment
* Participants with known prolongation of QT interval, ventricular cardiac arrhythmia, including torsades de pointes.
* Participants with ongoing proarrhythmic conditions such as uncorrected hypokalemia or hypomagnesemia, clinically significant bradycardia
* Participants with ongoing mononucleosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2027-11-06 (Estimated); Study Completion 2027-11-06 (Estimated)

PRIMARY OUTCOMES:
Percent of participants diagnosed with Helicobacter pylori using PYTEST® breath test at baseline | Baseline
  This measure determines the percent of participants who test positive for Helicobacter pylori at baseline. This is done using the PYTEST® 14C-Urea Breath Test. Participants will receive a diagnosis on-site, approximately 30 minutes after administration of urea capsule. This will allow immediate treatment free of charge (VOQUEZNA® Triple Pak®) initiation for positive eligible participants.

CONTACTS AND LOCATIONS:
Overall Officials: Shria Kumar, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No